CLINICAL TRIAL: NCT06503666
Title: Zambian Informed Motivated Aware Responsible Adolescent Girls and Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: University of Illinois at Chicago (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZAIMARA
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Implementation Science; Adolescent Girls and Young Adults; Low and Middle-Income Country
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: AGYW-MF will be randomized to either ZAIMARA or Health Promotion.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, masking of AGYW-MF participants is not possible. Our research assistants will be masked to the randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zambian Informed Motivated Aware Responsible Adolescent Girls and Young Adults(ZAIMARA) (Experimental): Intervention Arm
  Interventions: Behavioral: ZAIMARA
- Health Promotion (HP) (Experimental): Control Arm
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: ZAIMARA — The ZAIMARA curriculum focuses on strengthening communication between adolescent girls and young women (AGYW) and their mother figures (MF) to make healthy sexual decisions, to learn more about HIV, sexually transmitted infections (STIs), and pre-exposure prophylaxis (PrEP). The topics in the curriculum focus on effective communication, mothers talking to daughters on sex, HIV, STIs and PrEP. The intervention consists of participants attending a two day workshops with their MF.
  Other names:
  ZAIMARA
  Arms: Zambian Informed Motivated Aware Responsible Adolescent Girls and Young Adults(ZAIMARA)
Behavioral: Health Promotion — The health promotion (HP) curriculum focuses on healthy living by encouraging good nutrition, improving knowledge on violence recognition, management and support/resources, exercise, informed consumer behavior, alcohol and substance use.The intervention consists of participants attending a two day workshops with their MF.
  Other names:
  HP
  Arms: Health Promotion (HP)

SUMMARY:
The proposed hybrid effectiveness-implementation study will systematically adapt the Informed, Motivated, Aware, Responsible Adolescent Girls and Adults (IMARA) curriculum that was previously adapted for South Africa (IMARA-SA) to use in Zambia (will be renamed Zambian Informed, Motivated, Aware, Responsible Adolescent Girls and Adults (ZAIMARA) and evaluate the impact of ZAIMARA on improving adolescent girls and young women HIV testing, HIV and STI incidence, PrEP uptake and sexual risk behaviour. The study will also assess the impact of monthly mental health screening with referral versus a monthly nutrition and exercise screening on peer leaders job retention. We will also examine implementation factors and outcomes associated with ZAIMARA across five sites.

DETAILED DESCRIPTION:
The overall purpose of this study is to adapt the IMARA-SA curriculum for use in the Zambian context and test its impact on AGYW sexual behavior, as well as HIV and STI testing uptake and incidence, and PrEP uptake and persistence.

The study will be conducted in two phases. In Phase 1, we will systematically adapt IMARA-SA and the Health Promotion curriculum for use in the Zambian context using a combination of focus groups, CAB meetings, theater testing, and a formal pilot test. The IMARA curriculum focuses on strengthening communication between adolescent girls and young women (AGYW) and their mother figures (MF) to make healthy sexual decisions, to learn more about HIV, sexually transmitted infections (STIs), and pre-exposure prophylaxis (PrEP) while the health promotion (HP) curriculum promotes healthy living by encouraging good nutrition, knowledge on violence exercise, informed consumer behavior and substance use. The HP curriculum does not explicitly address HIV/STI prevention. Once adapted, the IMARA-SA will be renamed Zambian Informed, Motivated, Aware, Responsible Adolescent Girls and Adults (ZAIMARA).

In Phase 2 we will evaluate ZAIMARA's effectiveness on AGYW HIV testing, HIV and STI incidence, PrEP uptake, and sexual behavior. We will recruit 600 AGYW and MF dyads from the community with assistance from neighborhood health committee members (NHC). If participants agree to enroll in the study, consent/ assent will be obtained from AGYW and MF and they will be invited to participate in a 2-day workshop. On the first day of the workshop, the research assistants and study nurse will conduct clinical tests (HIV & STI), offer PrEP, collect baseline survey data, and randomize AGYW-MF to receive ZAIMARA or health promotion (HP). The peer leaders will administer the ZAIMARA and HP curriculum in the two days. Once the workshops are completed AGYW and MF dyads will graduate from the program and the study team will conduct follow-up assessments at 6, 12, 18, and 24 months. At the follow-up assessments, AGYW-MF will complete a survey, conduct clinical tests (HIV & STI), and receive PrEP (for eligible participants).

In addition to the trial component, will enroll the peer leaders who provide the intervention (ZAIMARA/HP) in the study. We aim to examine the impact of monthly mental health screening with referral versus a monthly nutrition and exercise screening on peer leader job retention. We will also evaluate ZAIMARA's feasibility, acceptability, appropriateness, fidelity, cost, and sustainability.

The study will occur in five geographically distinct catchment areas in Lusaka that feed into MoH district clinics/hospitals. The five Clinical Research Performance Sites (CRPS) are Kalingalinga Clinic, Chainda South Clinic, Chongwe Urban Clinic, Chelstone Clinic, and Matero first level hospital (subject to change if required). These clinics were selected based on the high volume of adolescents seeking services at these sites and the surrounding community population of AGYW that will allow us to enroll at least 2-3 AGYW-MF dyads per day in the respective sites.

ELIGIBILITY:
Inclusion Criteria:

Adolescent girls and young women (AGYW)

1. 15-19 years-old females (sex assigned at birth)
2. Unmarried
3. Residing outside the five study catchment areas
4. Speak Nyanja, Bemba, or English or a combination (the primary regional languages)
5. Willing and able to provide consent (> 18 years old) and/or assent (< 18 years old)
6. Not known to be living with HIV (i.e., no positive test and not on ART)

Mother Figures (MF)

1. selected to participate by the AGYW
2. if not the guardian/mother, agreed upon by the guardian/mother
3. > 24 years-old
4. living with or in daily contact with the AGYW
5. speak Nyanja, Bemba, or English or a combination
6. Willing and able to provide consent

Peer leaders (ZAIMARA & Health Promotion)

1. live in the community where they will be working
2. have prior experience working with young people
3. have a minimum grade 12 education
4. be proficient in reading and writing English and/or Nyanja or Bemba
5. are 22-29 years old for AGYW sessions
6. are >30 years-old for MF sessions

Exclusion Criteria:

AGYW

AGYW who are enrolled in other SRH interventions at the time of recruitment (to prevent confounding) or are known to be living with HIV (the needs of AGYW living with HIV are unique and not well-addressed in IMARA-SA, e.g., learning to disclose) will be excluded. Importantly, AGYW who test positive for HIV at the study's baseline assessment will be able to complete the workshops and referred for treatment to avoid stigma.

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All female participants (Sex assigned at birth for AGYW and MF)
Enrollment: 1200 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
AGYW HIV testing uptake | Within 6 months following delivery of ZAIMARA & HP curriculum
  Proportion of AGYW testing for HIV at 6 months

SECONDARY OUTCOMES:
Incident HIV infection and STIs, PrEP uptake, and AGYW sexual risk behavior | Within 6, 12, 18 and 24 months following delivery of ZAIMARA & HP curriculum
  Proportion of AGYW testing positive for HIV & STIs , Proportion requesting for PrEP and Proportion of AGYW engaging in sexual risk behaviour
AGYW HIV testing at 12, 18, and 24-months | Within 12, 18 and 24 months following delivery of ZAIMARA & HP curriculum
  Proportion of AGYW testing for HIV

CONTACTS AND LOCATIONS:
Locations (1):
- Chainda, Matero, Chelston, Chongwe and Kalingalinga, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
All necessary steps will be taken to ensure adherence to all NIH guidelines on sharing raw data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Pending
Access Criteria: Pending
URL: http://www.cidrz.org

REFERENCES:
- [Background] Donenberg GR, Wilson HW, Emerson E, Bryant FB. Holding the line with a watchful eye: the impact of perceived parental permissiveness and parental monitoring on risky sexual behavior among adolescents in psychiatric care. AIDS Educ Prev. 2002 Apr;14(2):138-57. doi: 10.1521/aeap.14.2.138.23899. PMID 12000232
- [Background] Donenberg GR, Emerson E, Bryant FB, Wilson H, Weber-Shifrin E. Understanding AIDS-risk behavior among adolescents in psychiatric care: links to psychopathology and peer relationships. J Am Acad Child Adolesc Psychiatry. 2001 Jun;40(6):642-53. doi: 10.1097/00004583-200106000-00008. PMID 11392341
- [Background] Donenberg G. Donenberg GR, Brown LK, Hadley W, Kapungu C, Lescano C. Family-based HIV-prevention program for adolescents with psychiatric disorders. In: Pequegnat W, Bell C, editors. Families and HIV/AIDS: Culture and contextual issues in prevention and treatment. New York: Springer; 2012.
- [Background] Donenberg G, Emerson E, Mackesy-Amiti ME, Fletcher F. Sexual risk among African American girls seeking psychiatric care: A social-personal framework. J Consult Clin Psychol. 2018 Jan;86(1):24-38. doi: 10.1037/ccp0000270. PMID 29300099
- [Background] Donenberg GR, Kendall AD, Emerson E, Fletcher FE, Bray BC, McCabe K. IMARA: A mother-daughter group randomized controlled trial to reduce sexually transmitted infections in Black/African-American adolescents. PLoS One. 2020 Nov 2;15(11):e0239650. doi: 10.1371/journal.pone.0239650. eCollection 2020. PMID 33137103
- [Derived] Donenberg GR, Sharma A, Kanguya T, Emerson E, Chhun N, Kasengele CT, Mweemba M, Mwenge M, Bosomprah S, Sissoko GD, Hosek S, Moore CB. A hybrid effectiveness implementation trial testing an HIV and STI prevention program for mother figures and their adolescent girls and young women delivered by peer leaders: ZAIMARA study protocol. BMC Public Health. 2025 Sep 30;25(1):3153. doi: 10.1186/s12889-025-24332-5. PMID 41029332